CLINICAL TRIAL: NCT07232979
Title: The Effectiveness of the Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) on Postoperative Analgesia and Recovery in Open-Heart Surgery: A Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: M-TAPA Block for Analgesia After Open-Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Collaborators: Emre ULUSOY (Unknown)
Responsible Party: Principal Investigator, eralp çevikkalp, assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 002
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Acute Pain
Keywords: M-TAPA block; Open-heart surgery; parasternal block; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Active Comparator): The M-TAPA and parasternal blocks will be administered before surgery.
  Interventions: Other: M TAPA block; Other: Parasternal blocks
- Group Control (Active Comparator): Preoperatively, a parasternal block and local anesthetic infiltration at the chest tube insertion sites will be administered to all patients.
  Interventions: Other: Parasternal blocks; Other: Local infiltration

INTERVENTIONS:
Other: M TAPA block — In the M-TAPA group, the block will be performed preoperatively with the patient in the supine position under ultrasound guidance using a high-frequency linear probe (GE ML6-15-D Matrix Linear, Boston, USA) and an 80-mm block needle (Stimuplex Ultra®, Braun, Melsungen, Germany). After identifying the appropriate plane between the transversus abdominis muscle and the lower surface of the costal cartilage, 5 mL of saline will be injected to confirm correct placement. Subsequently, 20 mL of 0.25% bupivacaine will be injected bilaterally (a total of 40 mL for both sides).
  Arms: Group M-TAPA
Other: Parasternal blocks — Before intubation, the block will be performed under aseptic conditions using a high-frequency ultrasound probe (GE ML6-15-D Matrix Linear, Boston, USA) placed immediately lateral to the sternum after identifying the second to fourth intercostal spaces. An 80-mm echogenic block needle (Stimuplex Ultra®, Braun, Melsungen, Germany) will then be advanced using an in-plane approach from the skin toward the plane between the pectoralis major and intercostal muscles. A total of 10 mL of 0.25% bupivacaine will be injected bilaterally.
Other: Local infiltration — Local anesthetic infiltration (10 mL of 0.25% bupivacaine) will be administered around the chest tube and mediastinal drain sites.
  Arms: Group Control

SUMMARY:
Postoperative pain following open-heart surgery is primarily caused by median sternotomy, although additional contributors include costovertebral joint stress related to sternal retraction and the presence of chest wall and mediastinal drains during the postoperative period. This pain is often severe, especially in the early postoperative hours, making effective management both challenging and essential. Insufficient pain control frequently necessitates high doses of opioids, which may lead to adverse effects such as nausea, vomiting, respiratory complications, and postoperative delirium. Excessive use of anesthetic agents or opioids can also delay extubation and prolong the process of weaning from mechanical ventilation.

The modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) is a regional anesthesia technique performed beneath the costal margin between the internal oblique and transversus abdominis muscles. It provides broad dermatomal coverage, extending approximately from the upper thoracic to the lower thoracic and upper lumbar segments. This study aims to evaluate the postoperative analgesic effectiveness of combining the M-TAPA block with a parasternal block in patients undergoing open-heart surgery.

DETAILED DESCRIPTION:
Postoperative pain following open-heart surgery is primarily caused by median sternotomy, although additional contributors include costovertebral joint stress related to sternal retraction and the presence of chest wall and mediastinal drains during the postoperative period. This pain is often severe, especially in the early postoperative hours, making effective management both challenging and essential. Insufficient pain control frequently necessitates high doses of opioids, which may lead to adverse effects such as nausea, vomiting, respiratory complications, and postoperative delirium. Excessive use of anesthetic agents or opioids can also delay extubation and prolong the process of weaning from mechanical ventilation.

The modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) is a regional anesthesia technique performed beneath the costal margin between the internal oblique and transversus abdominis muscles. It provides broad dermatomal coverage, extending approximately from the upper thoracic to the lower thoracic and upper lumbar segments. This study aims to evaluate the postoperative analgesic effectiveness of combining the M-TAPA block with a parasternal block in patients undergoing open-heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years with ASA physical status II-III who are scheduled to undergo elective open-heart surgery will be included.

Exclusion Criteria:

Patients who refuse to participate in the study

Patients with coagulopathy

Patients with a history of allergy or toxicity to local anesthetics

Patients with hepatic or renal failure

Patients with uncontrolled diabetes mellitus

Patients with uncontrolled hypertension

Mentally disabled patients

Patients receiving chronic pain therapy (opioid use)

Patients using antidepressant medications

Patients with neuropathic pain

Patients with infection at the injection site

Pregnant, suspected pregnant, or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 0, 2, 4, 8, 16 and 24 hours
  Fentanyl will be prepared at a concentration of 10 µg/mL, and patient-controlled analgesia (PCA) will be administered without a basal infusion, using a lock-out interval of 20 minutes and a bolus dose of 20 µg.

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | 0, 2, 4, 8, 16 and 24 hours
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
Global recovery scoring system (patient satisfaction scale)- QoR-15 | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  Researchers will use the Turkish version of the Quality Improvement Survey/QoR-15. PART A: Participants will be asked by researchers how they felt in the last 24 hours.(0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]) 1. Able to breathe easily 2. Been able to enjoy food 3. Feeling rested 4. Have had a good sleep 5. Able to look after personal toilet and hygiene unaided 6. Able to communicate with 7. Getting support from hospital doctors and nurses 8. Able to return to work or usual home activities 9. Feeling comfortable and in control 10. Having a feeling of general well-being PART B Participants will be asked by the researchers whether they have experienced any of the following in the last 24 hours. (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) 11. Moderate pain 12. Severe pain 13. Nausea or vomiting 14. Feeling worried or anxious 15. Feeling sad or depressed

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Dost B, De Cassai A, Balzani E, Tulgar S, Ahiskalioglu A. Effects of ultrasound-guided regional anesthesia in cardiac surgery: a systematic review and network meta-analysis. BMC Anesthesiol. 2022 Dec 29;22(1):409. doi: 10.1186/s12871-022-01952-7. PMID 36581838